CLINICAL TRIAL: NCT05231876
Title: Registre Wilson France
Brief Title: French Wilson Disease Registry
Acronym: WIL-FR
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CD/EB_19-003_APS
Record Dates: First submitted 2022-02-04; First posted 2022-02-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-06

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Recording of pathology-related information on the Wilson Register — Age, gender, date of diagnosis, clinical symptoms, ethnic charateristics and family tree will be collected and recorded on the Wilson Register during routine clinical care

SUMMARY:
This registry concerns adults and children with Wilson's disease. The collection of a large amount of data will allow a better understanding of the epidemiology of this rare disease, in particular the age of onset according to the hepatic or hepato-neurological forms, but also the geographical distribution of patients consulting in France. This database will also make it possible to know all the therapies prescribed to "Wilsonian" patients. The genetic study of these patients will make it possible to specify the various genetic mutations involved in Wilson's disease. The information (clinical, biological, radiological and genetic) relating to the disease will be entered by a doctor or a professional specialising in Wilson's disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from Wilson disease

Exclusion Criteria:

* Lack of written consent from the patient or their legal representative

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients suffering from Wilson disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Recording of pathology-related information on the Wilson Register | 1 hour
  The patient's age, sex, date of diagnosis, clinical symptoms, family tree and ethnic characteristics are collected by a physician or professional specialising in Wilson's disease during a routine care consultation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Wilson France Register — https://www.crmrwilson.com/registres/